CLINICAL TRIAL: NCT00604643
Title: Compassionate Use of the TALENT Aortic Cuff in the Treatment of Patients Previously Treated With the AneuRx Stent Graft System With Sub-Optimal Stent Graft Outcomes
Brief Title: Talent Aortic Cuff Stent Graft System Compassionate Use Registry
Status: No longer available | Type: Expanded Access
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: Investigational Plan #025
Record Dates: First submitted 2007-12-21; First posted 2008-01-30 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Abdominal Aneurysm; Endovascular Aortic Repair (EVAR); Endovascular Stent Graft; Endograft
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

INTERVENTIONS:
Device: TALENT Aortic Cuff Abdominal Stent Graft — Endovascular Aneurysm Repair

SUMMARY:
An evaluation of the TALENT Aortic Cuff in patients with existing AneuRx stent grafts who have experienced sub-optimal stent graft outcomes and are not deemed suitable candidates for treatment with an AneuRx Aortic Cuff.

DETAILED DESCRIPTION:
The primary purpose of this registry is to provide an endovascular means of treatment for those patients experiencing a sub-optimal outcome related to the implanted AneuRx bifurcated stent graft and who are not deemed suitable candidates for treatment with an AneuRx Aortic Cuff. A sub-optimal outcome is defined as either a Type I or Type III endoleak and/or an inadequate seal zone (< 1 cm). For Registry purposes, a Type III endoleak will be defined as a proximal modular endoleak.

ELIGIBILITY:
Inclusion Criteria:

* Patient >= 18 years of age
* Patient has a serious disease or condition
* No generally acceptable alternative for treating patient is available
* Patient has had the AneuRx stent graft system implanted >= 30 days
* Patient has suboptimal outcome with the AneuRx stent graft system as evidenced by one or more of the following:
* Type I endoleak
* Type III endoleak (Proximal, modular)
* Loss of seal zone
* Proximal aortic neck diameter >= 14mm and <= 30mm
* Angle between axis of the suprarenal aorta and aneurysm neck is <= 60 degrees
* Patient is able and willing to be available for 12,24,26,48 and 60 months post-procedure

Exclusion Criteria:

* Patient is pregnant of lactating
* Arterial access cannot be crossed with a delivery system
* Excessive vessel tortuosity
* Excessive aortic calcification
* AneuRx stent graft system implanted within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medtronic CardioVascular, Study Director — Medtronic Cardiovascular
Locations (50):
- United States (50):
  - Baptist Hospital, Montgomery, Alabama
  - Kaiser, Oakland, California
  - O'Connor Hospital, San Jose, California
  - Kaiser Hayward, Union City, California
  - Penrose Healthcare, Colorado Springs, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Washington Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - JA Haley Veterans Hospital, Tampa, Florida
  - St. Joseph's Hospital, Atlanta, Georgia
  - Gwinnett Hospital, Lawrenceville, Georgia
  - LaGrange Memorial Hospital, La Grange, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Via Christi Regional Medical center, Wichita, Kansas
  - University of Kentucky medical Center, Lexington, Kentucky
  - Baptist Hospital, Louisville, Kentucky
  - Southwest Medical Center, Lafayette, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - University of Massachusetts, Worcester, Massachusetts
  - Bon Secours Cottage Health Center, Saint Clair Shores, Michigan
  - Lakeland Regional Medical Center, Saint Joseph, Michigan
  - St. Cloud Hospital, Saint Cloud, Minnesota
  - Health Easst St. Joseph's Hospital, Saint Paul, Minnesota
  - CV Surgical Clinic, Jackson, Mississippi
  - St. Dominic-Jackson, Jackson, Mississippi
  - Jeff Anderson Regional Medical Center, Meridian, Mississippi
  - St. Luke's, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - NMVA Healthcare, Albuquerque, New Mexico
  - St. Luke's Healthcare, Utica, New York
  - Mission Hospital, Asheville, North Carolina
  - The Sanger Clinic-Carolinas Medical, Charlotte, North Carolina
  - Kaiser Sunnyside, Clackamas, Oregon
  - Pinnacle Health Hospital, Harrisburg, Pennsylvania
  - Hahnemann Univeristy Hospital, Philadelphia, Pennsylvania
  - Graduate Hospital, Philadelphia, Pennsylvania
  - Providence Hospital, Columbia, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - North Central heart Institute, Sioux Falls, South Dakota
  - Harlingen Medical Center, Harlingen, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Houston Northwest Medical Center, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - Henrico Doctors' Hospital, Richmond, Virginia
  - St. Luke's medical Center, Milwaukee, Wisconsin